CLINICAL TRIAL: NCT05036525
Title: Evaluation of the Efficacy and Safety of a High Molecular Weight Native Hyaluronic Acid Gel (HANBIO BarriGel) in Adhesion Prevention After Open Thyroidectomy: a Prospective, Randomized Controlled, Single Blind Study.
Brief Title: Evaluation of the Efficacy and Safety of a Hyaluronic Acid Gel in Adhesion Prevention After Open Thyroidectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HAN Biomedical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HAN2013001-CT02
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Adhesion; Thyroid Diseases
MeSH Terms: conditions — Tissue Adhesions; Thyroid Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- use HANBIO BarriGel (Experimental)
  Interventions: Device: HANBIO BarriGel
- No anti-adhesive product (No Intervention)

INTERVENTIONS:
Device: HANBIO BarriGel — an anti-adhesive product
  Arms: use HANBIO BarriGel

SUMMARY:
The aim of this study is to assess the safety and efficacy of HANBIO BarriGel to prevent thyroidectomy postoperative adhesions

DETAILED DESCRIPTION:
The objective of this study is to evaluate the efficacy of HANBIO BarriGel in the prevention of postoperative adhesion for patients who will undergo open thyroidectomy. The dysphagia and adhesion severity will be assessed at specific visits pre and/or post-operation for both treatment group and control group. The post-operative condition, and the adverse event information will be collected for evaluation of tolerability and safety of the product.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between 20 and 70 years of age.
* Patients diagnosed with benign goiter or thyroid cancer that will undergo open thyroidectomy (either unilateral or bilateral total thyroidectomy with or without central lymph node dissection).
* Naïve patients to thyroid surgery.
* Subjects are willing to comply with all aspects of the study and have signed informed consent form.

Exclusion Criteria:

* Pregnant or lactating female patients.
* Presence of severe and uncontrolled illness such as stroke, hypertension, diabetes, chronic renal failure, coagulopathy, drug abuse.
* Patients with previous neck radiotherapy within 1 year.
* Concurrent diseases/conditions which will be unable to evaluate the outcomes.
* Patients receiving any adhesion prevention adjuvant.
* Previous history of Keloid or hypertrophic scar.
* Anticoagulant used within a week from surgery.
* Subjects are hypersensitive to sodium hyaluronate.
* Participate in another clinical trial within 1 month.
* Patients presence of surgical site infection.
* Patients are with abnormal clinical test (appendix 1) result within one month or ECOG performance status (appendix 2) score ranged from 3-4.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Dysphagia Handicap Index (DHI) | Preoperative 6 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Keelung Chang Gung Memorial Hospital, Keelung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei